CLINICAL TRIAL: NCT04397692
Title: Inhaled NO for the Treatment of COVID-19 Caused by SARS-CoV-2 (US Trial)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: BAI_COV19_01_US
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Corona Virus Infection; COVID-19; SARS-CoV 2; Nitric Oxide; Respiratory Disease; Pneumonia, Viral; Inhaled Nitric Oxide
Keywords: COVID-19; Coronavirus; Inhaled Nitric Oxide; iNO; SARS-coronavirus; Virus
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Respiration Disorders; Pneumonia, Viral; Severe Acute Respiratory Syndrome; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Inhaled NO delivered using LungFit™ in addition to SST (Experimental): Patients will receive 80 ppm iNO for 40 min 4 times a day using LungFit™ device in addition to the standard of care.
  Interventions: Device: Nitric Oxide delivered via LungFit™ system
- Standard of care (No Intervention): Control - Standard of care

INTERVENTIONS:
Device: Nitric Oxide delivered via LungFit™ system — Patients will receive inhalations of 80 ppm for 40 min 4 times a day
  Arms: Inhaled NO delivered using LungFit™ in addition to SST

SUMMARY:
The purpose of this open label, randomized, study is to obtain information on the safety and efficacy of 80 ppm Nitric Oxide given in addition to the standard of care of patients with COVID-19 caused by SARS-CoV-2.

DETAILED DESCRIPTION:
Nitric Oxide (NO) is a small endogenously produced molecule recognized to play a critical role in the function of several body systems including the vasodilatation of smooth muscle, neurotransmission, regulation of wound healing and inhibition of pathogens. In-vitro studies have shown that NO inhibits the replication cycle of the severe acute respiratory syndrome coronavirus (SARS CoV) in vitro. The suggested mechanisms of actions of NO on SARS are an effect on the fusion between the S protein and its cognate receptor, ACE2, and reduction in viral RNA production in the early steps of viral replication. The primary aim of this feasibility study is to investigate the safety of intermittent NO, delivered via inhalation, in hospitalized patients with COVID-19. The primary endpoint in the study will be time to deterioration of respiratory symptoms determined by escalation to either non-invasive ventilation (NIV), high-flow nasal cannula (HFNC), or intubation.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 24 hours of hospital admission of patients diagnosed with COVID-19
* Patients with oxygen saturation less than 93 % on room air
* Shortness of breath, with symptom onset within the previous 8 days.
* Female subjects of childbearing potential should take adequate measures to avoid pregnancy
* Signed informed consent by the subject

Exclusion Criteria:

* Patients who are treated with or require high flow nasal cannula, CPAP, intubation, mechanical ventilation, or tracheostomy
* Diagnosis of acute respiratory distress syndrome
* Subjects diagnosed with immunodeficiency, with history of congestive or unstable heart disease, left ventricular dysfunction or myocardial damage, severe pulmonary hypertension and/or unstable hypertension
* Patients receiving drugs that have contraindications with NO.
* Breastfeeding or pregnancy as evidenced by a positive pregnancy test.
* Patients with active pulmonary malignancy or lung transplant
* Patients with a history of frequent epistaxis or significant hemoptysis

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Time to deterioration | 14 Days
  Time to deterioration measured by need for NIV, HFNC or intubation

SECONDARY OUTCOMES:
Time to NIV | 14 Days
  Time to non-invasive ventilation
Time to HFNC | 14 Days
  Time to high flow nasal cannula
Time to intubation | 14 days
  Time to intubation
Time to patient having stable oxygen saturation (SpO2) of greater than or equal to 93% | 14 days
  Time to patient having stable oxygen saturation (SpO2) of greater than or equal to 93%

OTHER OUTCOMES:
Need for supplemental oxygen | 14 days
  Need for supplemental oxygen
Change in viral load | 30 days
  Change in viral load
Duration of the Hospital Length of Stay (LOS) | 14 days
  Duration of the Hospital Length of Stay (LOS)
Mortality rate at Day 30 | 30 days
  Mortality rate at Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Ashik Tal, MD, Study Director — Beyond Air
Locations (1):
- Baptist Health Center for Clinical Research, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No